CLINICAL TRIAL: NCT04594642
Title: A Multicenter, Phase 1, Open-label, Dose-escalation and Expansion Study of AZD0486, a Bispecific Antibody Targeting CD19 in Subjects With B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study of AZD0486 in Subjects With B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7400C00006
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: B-cell Non Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Follicular Lymphoma
Keywords: NHL; DLBCL; HGBL; CD19; FL
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Adult subjects with B-NHL who will be enrolled into cohorts of incrementally increasing doses. Escalation is dependent upon ongoing review of emerging data by the Safety Monitoring Group (SMG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD0486 Monotherapy Dose Escalation in Subjects with B-NHL (Experimental): AZD0486 monotherapy will be administered intravenously on day 1 and 15 of 28 day cycles for a maximum of 2 years or until discontinuation criteria are met. Depending on cohort, subjects may receive priming or step-up dosing administered weekly during cycle 1 before reaching the target dose. Additional cohorts may be opened where subjects receive weekly dosing during Cycles 1-2. While on study, subjects will be monitored for safety and efficacy with periodic disease assessment with PET/CT. If subject achieves two consecutive CRs after completing C6, then they may be eligible for monthly dosing
  Interventions: Drug: AZD0486 IV

INTERVENTIONS:
Drug: AZD0486 IV — AZD0486 is a bispecific antibody targeting CD19 on tumor cells and CD3 on T-cells leading to T cell-mediated cytotoxicity of malignant B cells
  Other Names: TNB-486

SUMMARY:
This phase 1 study will investigate the safety, tolerability, pharmacokinetic, pharmacodynamic, and clinical activity of AZD0486, a CD19 x CD3 T-cell engaging bispecific antibody, in subjects with B-cell non-Hodgkin lymphoma (B-NHL).

DETAILED DESCRIPTION:
This dose escalation and optimization study, is evaluating the safety, tolerability, PK, PD and clinical activity of AZD0486 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven B-NHL, including DLBCL, HGBL, or FL.
* Relapsed/refractory cohorts:

In order to be eligible subjects must have received at least 2 prior lines of therapy and not be candidates for treatment regimens known to provide clinical benefit in B-NHL. CAR T-naive subjects are allowed if they have declined, are considered ineligible for, or do not have timely access to CAR T cell therapies.

* 1L FL cohorts: Subject has biopsy-proven FL Grade 1-3a per WHO 2016 classification, Stage II-IV, FL International Prognostic Index 2-5 that has not been treated with prior systemic lymphoma-directed therapy and requires initiation of treatment based on GELF criteria. Radiation to localized disease prior to study entry is allowed if >14 days from first dose.
* All Cohorts:

Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.

* Subject must have adequate liver, bone marrow and kidney function (eGFR ≥ 50 mL/min).
* Subject must have locally confirmed CD19 positivity (must be documented after time of progression from last CD19-targeted therapy, if received)
* Subject must have at least 1 measurable disease site
* Subject must have ANC >/= 1000/mm3, platelets >/= 50,000 mm3, hemoglobin >/= 8.0 g/dL. Transfusion and/or growth factor are allowed but counts must be stable for at least 72 hours afterwards prior to screening
* Subject must have a total bilirubin <1.5x ULN, AST/ALT < 3xULN

Exclusion Criteria:

* Subject has been diagnosed with or treated for another malignancy whose natural history or treatment may interfere with the safety or efficacy assessment of the investigational regimen.
* Subject has active central nervous system (CNS) involvement by their B-NHL. --Subjects may be eligible with a distant history of CNS involvement that has been adequately treated with no evidence of recurrence within last 6 months from screening.
* Subject has a history of leukemic presentation of their B-NHL (>5,000 circulating lymphoma cells/uL in the peripheral blood).
* Subject has history or presence of clinically significant CNS pathology
* Subject has CNS involvement from active or history of autoimmune disease.
* Subject received CD19 CAR T therapy within 3 months prior to first dose.
* Subject experienced Grade ≥ 3 cytokine release syndrome (CRS) following prior T-cell engager (TCE) or CAR T-cell therapy.
* Subject experienced Grade ≥ 2 neurotoxicity/immune effector cell-associated neurotoxicity syndrome (ICANS) following prior TCE or CAR T-cell therapy.
* Subject has received a peripheral autologous stem cell transplant (SCT) within 12 weeks, or an allogeneic SCT within 1 year of the first dose of study drug treatment or has received an SCT and requires ongoing immunosuppressive therapy.
* Subjects with human immunodeficiency virus (HIV) infection, or subjects with chronic or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV). HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Subjects with chronic HBV may be enrolled if the HBV viral load is undetectable on suppressive therapy, or if the subject has a documented cure. Subjects with HCV who have a documented cure may be enrolled.
* Subject has a history of major cardiac abnormalities.
* If female, subject must not be pregnant or breastfeeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2028-04-19 (Estimated); Study Completion 2028-04-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of subjects with Dose-limiting toxicities (DLT) | 28 days
  A DLT is defined as a TEAE that is not unequivocally due to the subject's underlying malignancy or other extraneous cause. DLT evaluable subjects are defined as those subjects who receive either the target dose of AZD0486 or priming dose(s) in any step-up dose schedule and are assessed for toxicities for the 28-day evaluation period.
  The NCI-CTCAE version 5.0 will be used (except for CRS and NT). A DLT will be evaluated as Non-hematologic, Hematologic, Cytokine Release Syndrome (CRS), or neurotoxicity.
Incidence of subjects with adverse events (AEs) and/or serious adverse events (SAEs) | From screening until 90 Days after end of treatment
  The incidence, timing, seriousness, and relationship to study treatment of adverse events will be evaluated.
Maximum Observed Serum Concentration of AZD0486 (Cmax) | 4 Weeks
  The maximum observed serum concentration on a concentration time curve.
Area under the concentration versus time curve from time zero to the last quantifiable time point prior to the next dose (AUClast) | 4 Weeks
  Area under the serum concentration-time curve from time zero to time of last measurable concentration.
Apparent terminal half-life (t1/2) of AZD0486 | From screening until 90 Days after end of treatment
  Terminal half-life (t1/2,) will be determined after infusion in Cycle 1 using non-compartmental methods.

SECONDARY OUTCOMES:
Anti-Lymphoma Activity by Objective Response Rate (ORR) | 48 months
  Objective response rate is defined as the proportion of subjects with a confirmed partial or complete response to treatment
Anti-Lymphoma Activity by Progression-Free Survival (PFS) | 48 months
  Progression-free survival time is defined as the time from the first dose of AZD0486 to progression or death, whichever occurs first
Anti-Lymphoma Activity by Duration of Objective Response (DOR) | 48 months
  The duration of objective response for a subject is defined as the time from the initial objective response to disease progression or death, whichever occurs first
Anti-Lymphoma Activity by Clinical Benefit Rate | 48 months
  Clinical benefit rate is defined as the proportion of subjects with a confirmed complete response, partial response or minor response, or stable disease for at least 24 weeks after responding to treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Sermer, MD, Study Director — AstraZeneca
Locations (23):
- United States (10):
  - Research Site, Tampa, Florida
  - Research Site, Louisville, Kentucky
  - Research Site, New Brunswick, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (4):
  - Research Site, Bedford Park
  - Research Site, Heidelberg
  - Research Site, Hobart
  - Research Site, Melbourne
- Japan (4):
  - Research Site, Chūōku
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Yamagata
- Research Site, Seoul, South Korea
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Kweishan
  - Research Site, Tainan
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
  Supporting
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Access Criteria:
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home